CLINICAL TRIAL: NCT05224284
Title: Impact of Blood and Ejaculate Bisphenol A Concentrations on ICSI Cycles Outcome in Patients With Male Factor
Brief Title: BPA Levels Relationship With IVF/ICSI Outcomes in Patients With Male Factor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor, Principal Investigator, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/21
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Male; IVF
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPA level (Other): BPA (Bisfenol A) in blood and ejaculate samples
  Interventions: Other: BPA levels

INTERVENTIONS:
Other: BPA levels — BPA (Bisfenol A) in blood and ejaculate samples

SUMMARY:
Association between blood and semen BPA levels and ICSI outcomes in patients with male factor

ELIGIBILITY:
Inclusion Criteria:

* female patients aged 23-40 years who underwent IVF due to male factor
* men with semen sample obtained from ejaculate
* male patients provided blood, and ejaculate samples on the oocyte retrieval day
* patients who did not smoke or use alcohol
* patients did not work in the plastic industry

Exclusion Criteria:

* men with a diagnosis of azoospermia
* patients who underwent IVF due to low ovarian reserve or unexplained infertility indications
* patients diagnosed with endometriosis
* patients with freeze-all cycles
* women with metabolic disease (such as hypertension or diabetes mellitus)
* patients (male or females) with a known genetic problem (male or female)

Ages: 23 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Exposure to BPA | 6 month
  Concentrations of Bisphenol A (BPA) will be quantified in the blood plasma, and ejaculate (individual and pooled samples) by use of ELİSA test in women with male factor

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)